CLINICAL TRIAL: NCT05155592
Title: Study of TNF-α Inhibitor Reduction or Discontinuation in Patients With Non-infectious Uveitis
Brief Title: Reduction or Discontinuation of TNF-α Inhibitor in Non-infectious Uveitis Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dan Liang (Other)
Responsible Party: Sponsor-Investigator, Dan Liang, PhD, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-ADA-Stop
Record Dates: First submitted 2021-12-09; First posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Uveitis; Adalimumab
Keywords: Uveitis; Adalimumab; TNF-α inhibitor
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with inactive uveitis (Experimental): Patients with non-infectious uveitis whose inflammation reached remission for at least six months after treatment with Adalimumab
  Interventions: Biological: reduction or discontinuation of Adalimumab

INTERVENTIONS:
Biological: reduction or discontinuation of Adalimumab — For patients with non-infectious uveitis whose inflammation stabilizes after treated with Adalimumab, extended dosing intervals to once a month, during which inflammatory status is monitored. If there was no recurrence within 6 months, Adalimumab was discontinued, and whether inflammation recurred after withdrawal was observed.

SUMMARY:
TNF-α inhibitors, like Adalimumab, have good efficacy in non-infectious uveitis, but long-term use can increase the risk of drugs, and the patient's financial burden is large. The objective of this study was to explore the reduction or withdrawal of Adalimumab in uveitis patients with stable drug control, and to evaluate the efficacy and safety of drug reduction in uveitis patients, as well as the impact on their vision prognosis.

DETAILED DESCRIPTION:
TNF-α inhibitors, like Adalimumab, have good efficacy in non-infectious uveitis, but long-term use will increase the risk of drugs, and the patient's financial burden is large. Previous studies have reported that tapering or discontinuation of Adalimumab may be considered in patients with stable disease. In clinical practice, some important questions about the feasibility of dose reduction in individual patients and the withdrawal plan remain unanswered. The objective of this study was to explore the reduction or withdrawal of Adalimumab in uveitis patients with stable drug control, and to evaluate the efficacy and safety of drug reduction in uveitis patients, as well as the impact on their vision prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of non-infectious uveitis
* nflammation was controlled for 6 months after drug remission was achieved using Adalimumab in combination with immunosuppressant therapy
* Family members and patients who are willing to stop should agree and accept relevant examinations
* The informed consent is read and signed by the patient or a legally authorized represent

Exclusion Criteria:

* Unwilling to sign informed consent
* There is systemic autoimmune disease uncontrolled situation
* Patients who may require surgery in the near future
* Vision meets the standards of low vision and blindness
* Silicone oil or gas filling after vitreous surgery

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
relapse rate of inflammation | 24 months
  The proportion of the number of uveitis relapse patients during the process of reduction or discontinuation

SECONDARY OUTCOMES:
Best corrected visual Acuity | 24 months
  increase of BCVA
macular structure | 24 months
  Macular thickness (MT). increase of central foveal thickness

CONTACTS AND LOCATIONS:
Overall Officials: Dan Liang, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yuan PD, Hu YW, Chen XQ, Chen GY, Pan Y, Lao HY, Liang D. Adalimumab Dose Reduction and Withdrawal in Stable Non-Infectious Pediatric Uveitis: An Open-Label, Prospective, Pilot Study. Ocul Immunol Inflamm. 2025 Apr;33(3):332-339. doi: 10.1080/09273948.2024.2343084. Epub 2024 Apr 23. PMID 38652891
- [Derived] Teabagy S, Wood E, Bilsbury E, Doherty S, Janardhana P, Lee DJ. Ocular immunosuppressive microenvironment and novel drug delivery for control of uveitis. Adv Drug Deliv Rev. 2023 Jul;198:114869. doi: 10.1016/j.addr.2023.114869. Epub 2023 May 10. PMID 37172782